CLINICAL TRIAL: NCT05977712
Title: Circadian Rhythm and Other Individual Factors Among Memory Clinic Patients
Brief Title: Circadian Rhythm and Other Factors in Memory Clinic Patients
Acronym: CIRCAME
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Fondation Rothschild Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230740; 2023-A01469-36 (Other: ID-RCB number)
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Dementia
Keywords: Circadian rhythm; Sleep disturbance; APOE; Retinal measures; Dementia subtypes, stages and progression; Alzheimer's disease; Lewy body dementia; Plasma biomarkers; Cerebrospinal fluid biomarkers; Individual risk factors; audiological function
MeSH Terms: conditions — Dementia; Parasomnias; Disease Progression; Alzheimer Disease; Lewy Body Disease | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CIRCAME: This is the full cohort of patients that compose the CIRCAME study (N estimated = 1500)
  Interventions: Other: Questionnaire; Other: Clinical examination; Other: Accelerometer port
- CIRCAME-EYE ancillary study: Patients from CIRCAME seen at the Fernand-Widal hospital who will also undergo an eye examination (CIRCAME-EYE, N estimated = 1100, a sub-group of CIRCAME)
  Interventions: Other: Eye examination
- CIRCAME-EAR ancillary study: Patients from CIRCAME seen at the Fernand-Widal hospital who will also undergo an audiolological examination (CIRCAME-EAR, N estimated = 1100, a sub-group of CIRCAME)
  Interventions: Other: Ear Examination

INTERVENTIONS:
Other: Questionnaire — The questionnaire includes information on socio-demographics (age, sex, education, occupation, marital status), behavioural (smoking, alcohol consumption, social functioning), and health-related factors (morbidities, treatment, sleep disturbance, eye diseases, frailty, falls).
  Groups: CIRCAME
Other: Clinical examination — This includes earing test, cognitive tests (mini-mental status examination, MemScreen), body mass index, waist circumference, blood pressure and blood tests (biomarkers of Alzheimer's disease, neurodegeneration, and other dementias).
  Groups: CIRCAME
Other: Accelerometer port — Participants will be wearing an accelerometer for 9 days.
  Groups: CIRCAME
Other: Eye examination — Eye fundus photo, OCT and OCT-A exams
  Groups: CIRCAME-EYE ancillary study
Other: Ear Examination — Otoscopic examination, Wideband tympanometry, Pure-tone and speech audiometry (in quiet and in noise), Auditory evoked potentials, Electroencephalogram with auditory stimulation
  Groups: CIRCAME-EAR ancillary study

SUMMARY:
The CIRCAME study is a bicentric study of patients from 2 memory clinics in Paris. The main objective is to identify circadian rhythm components and other individual risk factors (sociodemographic, behavioral, and health related factors) associated with the diagnosis of subtypes (AD, Lewy bodies, vascular, frontotemporal dementia) and stages (cognitively healthy, mild cognitive impairment, clinical dementia) of dementia, independent of known risk factors (sociodemographic and genetic) and assess the relevance of use of these factors in primary care for screen of dementia including subtypes and stages. A secondary objective is to determine factors associated with progression of the disease, in terms of cognitive decline and limitations in activities of daily living, as well as progression to dementia among cognitively healthy controls and patients with mild cognitive impairment, up to 15 years after the inclusion period.

DETAILED DESCRIPTION:
The diagnosis of Alzheimer's disease and other related dementias is mainly based on assessment of cognitive, behavioral and neuropsychological symptoms, functional limitations and imaging data/cerebrospinal fluid (CSF) biomarkers in some cases. These measures are primarily used in specialized clinics leading to a potential large number of dementia cases not being diagnosed. With population ageing, the number of people living with dementia is increasing and there is an urgent need for cost-effective, scalable tool for early, accurate screening of dementia cases, including both AD and other types of dementia, in primary care. Furthermore, the factors associated with the progression of the different types of dementia are still poorly understood, limiting the prospects for intervention to improve the quality of life of patients and their caregivers and to slow the progression of the disease.

This project aims to identify circadian rhythm components and other individual risk factors that could be used in primary care for dementia diagnosis (including its subtypes: AD, Lewy bodies, vascular, frontotemporal dementia) and stages (cognitively healthy, mild cognitive impairment, clinical dementia). A secondary objective is to determine factors associated with progression of the disease, in terms of cognitive decline and limitations in activities of daily living, as well as progression to dementia among cognitively healthy controls and patients with mild cognitive impairment.

This will be achieved using data from 1500 patients from 2 memory clinics in Paris from who data on sociodemographic, behavioral, and health related factors (such as reported sleep disturbance, plasma biomarkers, retina measures (in a subsample, CIRCAME-EYE) and audiological parameters (CIRCAME-Ear substudy)) will be measured at inclusion interview. Baseline examination will also include a wrist-mounted device for a measure of circadian rhythm and its related behaviors (physical activity and sleep), for which disruptions are thought to characterize dementia subtypes and stages. Information on dementia diagnosis and stages will come from memory clinic routine visits at the time of the inclusion; they will include subtypes (AD, Lewy bodies, vascular, frontotemporal dementia), cognitive stages (cognitively healthy, mild cognitive impairment, clinical dementia) and AD stages based on CSF biomarkers and clinical measures. Information on progression of the disease (change in cognitive function using the mini-mental status examination, change in limitations in activity of daily living) and incidence of dementia, institutionalization and mortality will be retrieved from patients' routine visits at memory clinics up to 15 years after the inclusion period.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age (18 or over)
* Signed informed consent form
* Patient affiliated to the french social security system

Exclusion Criteria:

* Skin allergy to plastic
* Diagnosis of psychiatric disorder that can explain all cognitive symptoms
* Inability to come accompanied for patients with a Mini-Mental State Examination (MMSE) cognitive score ≤18 or a clinician assessment indicating the need to be accompanied (e.g. wheelchair use, agitation)
* Participation at the time of inclusion and during the 9-day period of wearing the accelerometer in interventional research with potential impact on circadian rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1500 patients selected from two memory clinics in Paris (Lariboisière - F. Widal and Bretonneau).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2042-03 (Estimated)

PRIMARY OUTCOMES:
Dementia subtypes and stages (% at inclusion) | At inclusion
  Dementia subtypes and stages will be defined at inclusion based on the most recent routine visits at the memory center and categorised as: Alzheimer's disease, vascular dementia, Lewy body dementia, frontotemporal dementia), as having MCI (differentiating AD form of MCI and others), or being cognitively healthy.
  This consensus diagnosis of dementia subtypes among clinicians from the memory clinics is based on clinical examination consisting of a large battery of cognitive tests, assessment of behavioural and neuropsychological symptoms, and limitations in basic and instrumental activities of daily living (ADL/IADL), and additional examination of magnetic resonance imaging (MRI) and CSF biomarkers when AD is suspected or clinical symptoms do not provide an unequivocal diagnosis.
  This outcome will be examined as %
Dementia subtypes and stages (incidence) | From inclusion until last routine visit at the memory clinic within the 15 years following inclusion
  Dementia subtypes and stages will be defined on routine visits at the memory clini and categorised as: Alzheimer's disease, vascular dementia, Lewy body dementia, frontotemporal dementia), as having MCI (differentiating AD form of MCI and others), or being cognitively healthy.
  This consensus diagnosis of dementia subtypes among clinicians from the memory clinics is based on clinical examination consisting of a large battery of cognitive tests, assessment of behavioural and neuropsychological symptoms, and limitations in basic and instrumental activities of daily living (ADL/IADL), and additional examination of magnetic resonance imaging (MRI) and CSF biomarkers when AD is suspected or clinical symptoms do not provide an unequivocal diagnosis.
  This outcome will be examined among those with MCI and healthy controls as incident cases over time (up to 15 years after the inclusion) This outcome will be measured as part of the usual routine visits with the clinician (passive follow-up, vis
Alzheimer's disease stages (%) | At inclusion
  AD stages will be based on the most recent measure of CSF Aβ peptide level (Aβ42/40 ratio) to assess the A+ criterion, p-Tau 181 to assess the T+ criterion, and clinical examination to assess the CogFI+ criterion (cognitive impairment and/or neurobehavioural symptoms with functional impact on daily life). Patients will be categorised based on all combinations of positivity status on A, T and CogFI and % in each category will be compared.
  This analysis will be among those with CSF biomarkers measured as part of their routine visit at the memory clinics.
Alzheimer's disease stages (change in) | From inclusion until last routine visit at the memory clinic within the 15 years following inclusion
  AD stages change will be based on the most recent measure of CSF Aβ peptide level (Aβ42/40 ratio) to assess the A+ criterion, p-Tau 181 to assess the T+ criterion, and clinical examination to assess the CogFI+ criterion (cognitive impairment and/or neurobehavioural symptoms with functional impact on daily life). Patients will be categorised based on all combinations of positivity status on A, T and CogFI and change in categories since inclusion status will be compared.
  This analysis will be among those with CSF biomarkers measured as part of their routine visit at the memory clinics.
  This outcome will be measured as part of the usual routine visits with the clinician (passive follow-up, visit not specific to CIRCAME)

SECONDARY OUTCOMES:
Level of Amyloid β 42/40 ratio (concentration) | At inclusion
  Amyloid β 42/40 ratio, a marker of AD pathology, will be measured based on Simoa 4-plex E assay of plasma sample from the inclusion visit
Level of neurofilament light (NfL) (concentration) | At inclusion
  Neurofilament light (NfL), a marker of neurodegeneration in all neurodegenerative diseases, will be measured based on Simoa 4-plex E assay of plasma sample from the inclusion visit
Level of Glial fibrillary acidic protein (GFAP) (concentration) | At inclusion
  Glial fibrillary acidic protein (GFAP), a marker of astrocytosis, will be measured based on Simoa 4-plex E assay of plasma sample from the inclusion visit
Level of phosphorylated tau (p-tau) (concentration) | At inclusion
  Phosphorylated tau (p-tau) for detection of early AD-related tauopathy and disease staging ,will be measured based on ALZ-path Simoa p-tau 217 assay of plasma sample from the inclusion visit
Level of baseline cognition (mini-mental status examination) | At inclusion
  At inclusion the mini-mental status examination will be assessed by trained nurse and with possible scores between 0 and 30
Change in cognitive performance (mini-mental status examination) | From inclusion until last routine visit at the memory clinic within the 15 years following inclusion
  The mini-mental status examination will be extracted from memory clinic records from routine visits with the clinician at memory clinics
Level of baseline cognition (MemScreen) | At inclusion
  At inclusion the MemScreen digital cognitive test will be assessed by trained nurse and with possible scores between 0 and 34
Change in cognitive performance (MemScreen) | From inclusion until last routine visit at the memory clinic within the 15 years following inclusion
  The MemScreen will be extracted from memory clinic records from routine visits with the clinician at memory clinics
Level of limitations in basic activities of daily living | At inclusion
  At inclusion the number of limitations in activities of daily living ((dressing, walking, bathing, eating, continence, using toilet) will be assessed by trained nurse and with possible scores between 0 and 6
Change in limitations in basic activities of daily living | From inclusion until last routine visit at the memory clinic within the 15 years following inclusion
  Change since inception in the number of limitations in activities of daily living (dressing, walking, bathing, eating, continence, using toilet) will be examined. The number of limitations in activities of daily living will be extracted from memory clinic records from routine visits with the clinician at memory clinics
Level of limitations in instrumental activities of daily living | At inclusion
  At inclusion the number of limitations in activities of daily living (cooking, shopping for grocery, telephone calls, taking medication, using transports, managing money) will be assessed by trained nurse and with possible scores between 0 and 6
Change in limitations in instrumental activities of daily living | From inclusion until last routine visit at the memory clinic within the 15 years following inclusion
  Change since inception in the number of limitations in instrumental activities of daily living (cooking, shopping for grocery, telephone calls, taking medication, using transports, managing money) will be examined. The number of limitations in instrumental activities of daily living will be extracted from memory clinic records from routine visits with the clinician at memory clinics.
Incidence of institutionalization | From inclusion until last routine visit at the memory clinic within the 15 years following inclusion
  Information on entrance in institution (medical institution for long stay) will come from memory clinics records.
Incidence of hospitalisation | From inclusion until last routine visit at the memory clinic within the 15 years following inclusion
  Information on entrance in hospitalisation (planned or unplanned) will come from memory clinics records.
Incidence of death | From inclusion until last routine visit at the memory clinic within the 15 years following inclusion
  Information on death (date) will come from memory clinics records.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de neurologie Cognitive / CMRR, Paris, France
  - Hôpital de Jour Gériatrique et consultation mémoire, Paris, France

IPD SHARING:
Plan to Share IPD: No